CLINICAL TRIAL: NCT06463275
Title: Determination of the 99th Percentile Upper Reference Limits (URLs) for the SpinChip High Sensitivity Cardiac Troponin I (SpinChip Hs-cTnI) Test
Brief Title: SpinChip Hs-cTnI Determination of the 99th Percentile URL
Acronym: HEAT-3
Status: Completed | Type: Observational
Sponsor: SpinChip Diagnostics ASA (Industry)
Collaborators: Aurevia (Industry); CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Design Protocol-03542; CIV-SE-23-12-045358 (Other: EUDAMED)
Record Dates: First submitted 2024-06-07; First posted 2024-06-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; High-sensitive; Point of Care; Troponin I; Near-patient test; Heart attack; 99th percentile upper reference limit
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Li-heparin plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SpinChip hs-cTnI — SpinChip Platform, consisting of the SpinChip hs-cTnI test (self-contained cartridge) and SpinChip Analyzer (instrument).

SUMMARY:
During a heart attack, the protein troponin I is released from the heart muscle into the bloodstream. Measurements of cardiac troponin in blood are used as an aid in the diagnosis of heart attack. Low levels of troponin are also present in the blood stream of healthy individuals and can be detected by high-sensitive troponin tests. The SpinChip hs-cTnI test is a new high-sensitive test for measuring the amount of cardiac troponin I in the bloodstream as an aid in the diagnosis of heart attack.

The purpose of this study is to determine the upper reference limits (URLs) for the SpinChip hs-cTnI test in a healthy population.

DETAILED DESCRIPTION:
Cardiac troponins are widely used as a biomarker to aid in the diagnosis of Acute myocardial infarction (AMI). These structural proteins are essential in regulating contraction in cardiac muscle cells, and they are sensitive and specific biochemical markers of myocardial damage.

During a heart attack, cardiac muscle cells are injured and release the cardiac marker troponin I (cTnI) into the bloodstream. High-sensitive troponin tests may detect the increase of cardiac troponin in blood within hours after the symptoms of a heart attack has started.

According to the European Society of Cardiology (ESC) 2023 guideline for acute coronary syndrome (ACS) in patients presenting without persistent ST-segment elevation, an elevated cTn value above the 99th percentile upper reference limit (URL) indicates myocardial injury, and when accompanied by evidence of acute myocardial ischemia, the disease is defined as AMI. The diagnostic threshold (99th percentile URL) for each hs-cTn test method must be specifically established.

The SpinChip high-sensitivity cardiac troponin I (hs-cTnI) test is a new high-sensitive test for measuring troponin I in blood samples, and the analysis may be performed close to the patient (near-patient test). The results may be obtained within 10 minutes, compared to approximately 1 hour for normal laboratory analysis using fresh venous whole blood and plasma samples.

The SpinChip Platform consists of the SpinChip hs-cTnI test and the SpinChip Analyzer and may be used at the emergency department to evaluate patients presenting with symptoms of acute myocardial infarction (chest pain). The test can use blood from finger prick or venous blood samples, either as whole blood or separated into plasma.

This study is a multicentre, prospective, observational, non-randomised, clinical performance study in healthy subjects to determine the 99th percentile URLs for the SpinChip hs-cTnI test according to recommendations from the International Federation of Clinical Chemistry and Laboratory Medicine (IFCC).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed written informed consent
* 18-80 years old
* Estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73 m2 for subjects 18-65 years and > 50 mL/min/1.73 m2 for subjects > 66 years
* Haemoglobin A1c (HbA1c) < 6.5% (< 48 mmol/mol)
* NT-proBNP (N-terminal prohormone of brain natriuretic peptide) < 125 ng/L or BNP (brain natriuretic peptide) < 35 ng/L

Exclusion Criteria:

* All known cardiovascular or cardiac diseases (evaluated using questionnaire; personal history of acute myocardial infarction (AMI) or other cardiac diseases (angina, stroke, atrial fibrillation, peripheral vascular disease (PVD), deep vein thrombosis (DVT), pulmonary embolism (PE), cardiac valve disease, heart failure)
* Treatment for hyperlipidaemia (medication reported in questionnaire)
* Hypertension (as judged by the investigator) or use of medication for hypertension (medication reported in questionnaire)
* Treatment for diabetes, including dietary treatment (reported in questionnaire)
* Abnormal BMI (body mass index) (< 18 kg/m2 or > 35 kg/m2), calculated from data collected during enrolment visit
* Current smokers (reported in questionnaire)
* Major illness or chronic disease that could affect the heart (lung, liver, unstable or nontreated thyroid disease, or autoimmune diseases (evaluated using questionnaire)
* History of cancer within the last 5 years (based on questionnaire) except basal cell carcinoma (in situ)
* Recent acute hospitalisation (within last 3 months, reported in questionnaire)
* Pregnancy (reported in questionnaire)
* Already included in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 800 healthy subjects with a balanced gender distribution (minimum 400 females and 400 males).
Sampling Method: Non-Probability Sample
Enrollment: 1355 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Overall 99th percentile URL | 1 day
  Determine the overall 99th percentile URL of the SpinChip hs-cTnI test using cTnI results obtained from analysis of Li-Heparin whole blood and Li-Heparin plasma samples using the non-parametric method

SECONDARY OUTCOMES:
Sex-specific 99th percentile URLs | 1 day
  Calculate the sex-specific 99th percentile URLs of the SpinChip hs-cTnI test using cTnI results obtained from analysis of Li-Heparin whole blood and Li-Heparin plasma samples using the non-parametric method.
Percentage of measurable values above LoD | 1 day
  To assess the sensitivity of the SpinChip hs-cTnI test quantified as the percentage (%) of measurable values (>limit of detection, LoD) for males, females, and the overall population, for each sample type (Li-Heparin whole blood and Li-Heparin plasma).
Incidence of AEs, ADEs, and DDs | 1 day
  Assess safety of the SpinChip Platform, as measured by adverse events (AEs), adverse device effects (ADEs) and device deficiencies (DDs).

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nilsson, MD/PhD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (4):
- Sweden (4):
  - Clinical Trial Consultants (CTC) GoCo, Mölndal, Gothenburg
  - CTC Clinical Trial Consultants AB, Uppsala, Uppsala County
  - Clinical Trial Consultants (CTC) Ebbepark, Linköping
  - Phase I-IV Research Unit Karolinska, Solna

IPD SHARING:
Plan to Share IPD: No